CLINICAL TRIAL: NCT00646321
Title: A 12 Week, Randomized, Double-Blind, Double-Dummy, Active-Controlled Study of SYMBICORT pMDI Administered Once Daily in Children and Adolescents 6 to 15 Years of Age With Asthma - SPROUT
Brief Title: Efficacy of Symbicort pMDI Administered Once Daily in Children and Adolescents During 12 Weeks - SPROUT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SD-039-0725; D5896C00725
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: asthma; children; adolescents; Symbicort; budesonide/ formoterol; budesonide
MeSH Terms: conditions — Asthma | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): budesonide/formoterol
  Interventions: Drug: budesonide/formoterol (Symbicort)
- 2 (Active Comparator): budesonide
  Interventions: Drug: budesonide

INTERVENTIONS:
Drug: budesonide/formoterol (Symbicort)
  Other Names: Symbicort
  Arms: 1
Drug: budesonide
  Arms: 2

SUMMARY:
The purpose of this study is to compare Symbicort with budesonide alone for the treatment of asthma in children aged 6 to 15 years

ELIGIBILITY:
Inclusion Criteria:

* At least 6 and maximally 15 years of age
* Diagnosis of asthma and baseline lung function tests as determined by the protocol
* Has required and received treatment with inhaled corticosteroids within the timeframe and doses specified in the protocol

Exclusion Criteria:

* Severe asthma
* Has required treatment with any non-inhaled corticosteroids within previous 4 weeks, has sensitivity to drugs specified in the protocol or requires treatment with beta-blockers

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 540 (Estimated)
Dates: Start 2003-04; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Change in evening PEF | Daily throughout the 12 week treatment period

SECONDARY OUTCOMES:
Lung function, asthma symptoms, use of rescue medication and parent/caregiver/physician reported outcomes | Daily throughout the 12 week treatment period
Routine safety assessments described in the protocol | 2-4 assessments within 12 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bonuccelli, Study Director — AstraZeneca

REFERENCES:
- [Derived] Eid NS, Noonan MJ, Chipps B, Parasuraman B, Miller CJ, O'Brien CD. Once- vs twice-daily budesonide/formoterol in 6- to 15-year-old patients with stable asthma. Pediatrics. 2010 Sep;126(3):e565-75. doi: 10.1542/peds.2009-2970. Epub 2010 Aug 16. PMID 20713475